CLINICAL TRIAL: NCT02613689
Title: Addressing Tobacco Use Disparities Through an Innovative Mobile Phone Intervention: The Text to Forgo Smokeless Tobacco
Brief Title: Addressing Tobacco Use Disparities Through an Innovative Mobile Phone Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063791; 1R15CA198841-01 (NIH)
Record Dates: First submitted 2015-11-12; First posted 2015-11-24 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Smokeless Tobacco Cessation
Keywords: smokeless tobacco, text message, tobacco cessation, tobacco
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use

ARMS (2):
- Scheduled Gradual Reduction (SGR) (Experimental): Subjects will receive the Scheduled Gradual Reduction (SGR) intervention, as well as SMS support text messages.
  Interventions: Behavioral: Scheduled Gradual Reduction (SGR); Behavioral: Text Messages
- Control Group (Active Comparator): Subjects will receive SMS support text messages
  Interventions: Behavioral: Text Messages

INTERVENTIONS:
Behavioral: Scheduled Gradual Reduction (SGR) — Participants in this group will group will receive the Scheduled Gradual Reduction (SGR) smokeless tobacco cessation reduction intervention via text message over a period of four weeks. Participants will initially report their smokeless tobacco use according to their usual habit, and over the course of the intervention be directed via text message precise times to start and stop each instance of smokeless tobacco use, gradually reducing the occurrences of use. In addition, this group will also receive the support messages that are sent to the control group.
  Arms: Scheduled Gradual Reduction (SGR)
Behavioral: Text Messages — Participants in this group will receive text messages about smokeless tobacco cessation in the form of counseling messages at various times throughout the day over a period of four weeks.

SUMMARY:
The purpose of this study is to evaluate the feasibility, acceptability and preliminary efficacy of a Scheduled Gradual Reduction (SGR) intervention via Short Message Service (SMS) text messaging plus SMS Support Messages in decreasing smokeless tobacco use in a rural population.

DETAILED DESCRIPTION:
Participants will be randomized to either the Scheduled Gradual Reduction (SGR) group or the control group. All participants in both groups will complete surveys at the baseline, end of program, and 6 month time points. All participants in both groups will also receive supportive counseling text messages at various times during the day over a period of 4 weeks.

Participants assigned to the SGR intervention group will receive their intervention, in addition to the supportive counseling messages received by the control group, via text message over a period of four weeks. Participants will initially report their smokeless tobacco use according to their usual habit, and over the course of the intervention be directed via text message precise times to start and stop each instance of smokeless tobacco use, gradually reducing the occurrences of use.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Have used smokeless tobacco for the last year, currently (past 30 days) uses smokeless tobacco daily, and use of at least one or more tins/cans per week
* Have an address in a rural census tract defined by a RUCA code of 4-10.
* Interested in participating in a cessation program
* Have access to a cell phone with unlimited texting ability and have knowledge of text messaging

Exclusion Criteria:

* Non-English speaking
* Have smoked cigarettes or used any other tobacco product in the past 30 days (i.e., dual user)
* Currently participating in a smokeless tobacco cessation study
* Family member participating in a smokeless tobacco cessation study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of Return Text Messages sent in Response to SGR Intervention | 1 month
  Assessed via text history
Proportion of Support Messages Read by Participants | 1 month
  Self-report
Ratings of Usefulness of the Intervention Received | 1 month
  Ratings will be assessed via patient questionnaire.
Quit Rate at 1 month | 1 month
  Quit rate will be assessed by participant self report via questionnaires. Participants will also be asked to provide a saliva sample to check for nicotine if they report that they have quit using smokeless tobacco.
Quit Rate at 6 Months | 6 months
  Quit rate will be assessed by participant self report via questionnaires. Participants will also be asked to provide a saliva sample to check for nicotine if they report that they have quit using smokeless tobacco.

CONTACTS AND LOCATIONS:
Overall Officials: Devon Noonan, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University School of Nursing, Durham, North Carolina, United States